CLINICAL TRIAL: NCT02038049
Title: A Randomized, Partially Blind, Placebo-controlled, Proof-of-concept Study to Assess the Effect of a Single Infusion of VAY736 on Disease Activity as Measured by Brain MRI Scans in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: A Study to Assess the Effect of a Single Infusion of VAY736 on Disease Activity in Patients With Relapsing-remitting Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study recruitment was terminated based on strategic considerations after 8 patients were enrolled.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736X2202; 2013-002324-16 (EudraCT Number)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-10

CONDITIONS: Relapse Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Magnetic Resonance Imaging; VAY736; Lanalumab; monoclonal antibody; gadolinium [Gd]-enhancing lesions; B-Cell
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAY736 (Experimental): Intravenous infusion of VAY736
  Interventions: Drug: VAY736
- Placebo to VAY736 (Placebo Comparator): Matching placebo (infusion bag) administered intravenously. Placebo randomized patients were offered optional VAY736 administration after week 16
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VAY736 — Single intravenous infusion of VAY736 (10 mg/kg)
  Other Names: Lanalumab
  Arms: VAY736
Drug: Placebo — Placebo to VAY736
  Arms: Placebo to VAY736

SUMMARY:
This was a randomized, partially blinded, placebo-controlled, non-confirmatory study to assess the effects of a single infusion of VAY736 on disease activity as measured by brain MRI scans in patients with relapsing-remitting multiple sclerosis (RRMS).

DETAILED DESCRIPTION:
The study was planned to be conducted in approximately 96 patients. However, after enrolling 8 patients, the recruitment was terminated based on strategic considerations.

ELIGIBILITY:
Key inclusion criteria:

* Male and female patients aged 18 to 55 years.
* Diagnosis of MS as defined by the 2010 revised McDonald criteria (Polman et al 2011).
* A relapsing-remitting course of disease with:

  * at least 1 documented relapse during the previous 12 months (but not within 30 days prior to randomization ), or
  * a positive Gd-enhancing lesion on brain MRI scan at screening.
* An Expanded Disability Status Scale (EDSS) score of 0-5.0 inclusive at screening.
* No evidence of a relapse within 30 days prior to randomization.

Key exclusion criteria:

* A manifestation of another type of MS other than RRMS.
* Findings on screening or baseline brain MRI inconsistent with the diagnosis of MS.
* History of chronic disease of the immune system other than MS, or a known immunodeficiency syndrome.
* Score "yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS, if this ideation occurred in the past 6 months, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), if this behavior occurred in the past 2 years.
* Women of child-bearing potential and Pregnant or nursing (lactating) women.
* Screening CBC (complete blood count) laboratory values as follows:
* Hemoglobin levels below 10.0 g/dL
* Total leukocyte count less than 3,000 cells/µL
* Neutropenia, defined as absolute neutrophil counts less than 1500 cells/mm3
* Platelets less than 100,000/µL

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2015-05-05 (Actual); Study Completion 2018-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (2):
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, San Diego, California
- Novartis Investigative Site, Hradec Králové, Czechia
- Ukraine (2):
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Lviv

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 5 centers in 3 countries: Czech Republic (1), Ukraine (2 sites) and USA (2 sites).
Pre-assignment Details: The study was planned to be conducted in approximately 96 patients. However, after enrolling 8 patients, the recruitment was terminated based on strategic considerations.
Period: Overall Study
Arm/Group | VAY736 | Placebo to VAY736
Started (All randomized patients were included in the Full Analysis (FAS) and Safety Set) | 4 | 4
Pharmacodynamic (PD) Analysis Set (At least one dose of study drug and one evaluable PD assessment) | 4 | 4
Completed | 3 | 4
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAY736 | Placebo to VAY736 | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.0 (10.42) | 42.0 (2.45) | 37.0 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 3 | 4 | 7
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of New T1-weighted Gadolinium (Gd)-Enhancing Lesions at Weeks 8, 12 and 16
Description: The effect of VAY736, compared to placebo on the cumulative number of new gadolinium [Gd]-enhancing lesions on T1-weighted brain MRI scans in relapsing-remitting multiple sclerosis (RRMS) patient population at weeks 8, 12 and 16. Only descriptive statistics performed.
Time Frame: Week 8, Week 12, Week 16
Population: Pharmacodynamic (PD) analysis set, which consisted of all patients who received at least one dose of study drug during the treatment and one evaluable PD assessment, was considered
Measure: Number; unit: Lesions
Arm/Group | VAY736 | Placebo to VAY736
Number analyzed (Participants) | 4 | 4
Lesions
  Week 8 | 5 | 1
  Week12 | 5 | 2
  Week 16 | 6 | 3

2. Secondary Outcome: Number of All T1-weighted Gadolinium (Gd)-Enhancing Lesions at Weeks 4, 8, 12 and 16
Description: Magnetic resonance imaging (MRI) scanning of the brain was performed at screening/baseline, week 4, week 8, week 12 and week 16 to assess all T1-weighted Gadolinium (Gd) enhancing lesions. Each MRI scan was reviewed by a local neuro-radiologist. Only descriptive statistics performed.
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Number; unit: Lesions
Arm/Group | VAY736 | Placebo to VAY736
Number analyzed (Participants) | 4 | 4
Lesions
  Week 4 | 19 | 2
  Week 8 | 20 | 2
  Week 12 | 20 | 3
  Week 16 | 21 | 4

3. Secondary Outcome: Number of New T1-weighted Gadolinium (Gd)-Enhancing Lesions at Weeks 4, 8, 12 and 16
Description: Magnetic resonance imaging (MRI) scanning of the brain was performed at screening/baseline, week 4, week 8, week 12 and week 16 to assess all new T1-weighted Gadolinium (Gd) enhancing lesions. Each MRI scan was reviewed by a local neuro-radiologist. Only descriptive statistics performed.
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Number; unit: Lesions
Arm/Group | VAY736 | Placebo to VAY736
Number analyzed (Participants) | 4 | 4
Lesions
  Week 4 | 4 | 1
  Week 8 | 1 | 0
  Week 12 | 0 | 1
  Week 16 | 1 | 1

4. Secondary Outcome: Number of New or Enlarging T2-weighted Gadolinium (Gd)-Enhancing Lesions at Weeks 4, 8, 12 and 16
Description: Magnetic resonance imaging (MRI) scanning of the brain was performed at screening/baseline, week 4, week 8, week 12 and week 16 to assess T2 hyperintense lesions (new or enlarging T2-weighted lesions). Each MRI scan was reviewed by a local neuro-radiologist. Only descriptive statistics performed.
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Number; unit: Lesions
Arm/Group | VAY736 | Placebo to VAY736
Number analyzed (Participants) | 4 | 4
Lesions
  Week 4 | 279 | 94
  Week 8 | 277 | 93
  Week 12 | 276 | 91
  Week 16 | 264 | 91

5. Secondary Outcome: T2 Burden of Disease (Total Volume of T2-weighted Lesions) at Weeks 4, 8, 12 and 16.
Description: Magnetic resonance imaging (MRI) scanning of the brain was performed at screening/baseline, week 4, week 8, week 12 and week 16 to assess T2 burden of disease. Each MRI scan was reviewed by a local neuro-radiologist. Only descriptive statistics performed.
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Number; unit: mm3 of T2-weighted lesions
Arm/Group | VAY736 | Placebo to VAY736
Number analyzed (Participants) | 4 | 4
mm3 of T2-weighted lesions
  Week 4 | 20108.9 | 17706
  Week 8 | 18998.9 | 16785
  Week 12 | 18484.1 | 15996
  Week 16 | 18102.7 | 17919

6. Secondary Outcome: Number of Subjects Without Any New MRI Disease Activity at Weeks 4, 8, 12 and 16.
Description: Magnetic resonance imaging (MRI) scanning of the brain was performed at screening/baseline, week 4, week 8, week 12 and week 16 to assess patients without any new MRI disease activity (no new Gd-enhancing lesions nor new or enlarging T2 lesions). Each MRI scan was reviewed by a local neuro-radiologist. Only descriptive statistics performed.
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VAY736 | Placebo to VAY736
Number analyzed (Participants) | 4 | 4
Participants
  Week 4 | 4 | 2
  Week 8 | 1 | 0
  Week 12 | 0 | 1
  Week 16 | 3 | 3

7. Secondary Outcome: Proportion of Relapse-free Patients Over the 16 Weeks of the Treatment Period.
Description: A relapse is defined as the appearance of a new neurological abnormality, or worsening of previously stable, or improving pre-existing neurological abnormality, separated by at least 30 days from the onset of a preceding clinical demyelinating event. The abnormality must be present for at least 24 hours and occur in the absence of fever (<37.5 C) or infection. A relapse was considered confirmed when confirmed by an Extended disability status scale (EDSS)-certified physician who was not involved in the treatment of the patient, was blinded to treatment allocation, and had no access to patient medical records. It was recommended that this occurs within 5 days of the onset of symptoms. A relapse was confirmed when it was accompanied by an increase of at least half a point (0.5) on the EDSS or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS). Only descriptive statistics performed.
Time Frame: Week 0 (Day 1), Week 4, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | VAY736 | Placebo to VAY736
Number analyzed (Participants) | 4 | 4
Participants
  Week 0 (Day 1): Relapse-free | 4 | 4
  Week 0 (Day 1): Relapse | 0 | 0
  Week 4: Relapse-free | 4 | 4
  Week 4: Relapse | 0 | 0
  Week 8: Relapse-free | 4 | 4
  Week 8: Relapse | 0 | 0
  Week 12: Relapse-free | 4 | 4
  Week 12: Relapse | 0 | 0
  Week 16: Relapse-free | 3 | 3
  Week 16: Relapse | 1 | 1

8. Secondary Outcome: Number of Participants With On-Treatment Adverse Events, Serious Adverse Event, and Death
Description: Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) to demonstrate that VAY736 is safe for the treatment of patients with relapsing-remitting multiple sclerosis through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive statistics performed.
Time Frame: From first dosing (single administration, Day 1) up to End of Study Visit (EOS) depending on B cell recovery (ranging from week 48 to 216)
Population: The Safety Set, which consisted of all patients who received at least one dose of study drug during the treatment period, was considered
Measure: Count of Participants; unit: Participants
Groups:
- VAY736 Administered at Visit 2 (Day 1): Intravenous infusion of VAY736 at Visit 2 (Day 1)
- VAY736 Administered at Visit 7 (Week 16 - Week 17): Intravenous infusion of VAY736 at Visit 7 (Week 16 - Week 17)
- Placebo Administered at Visit 2: Matching placebo (infusion bag) administered intravenously at Visit 2. Placebo randomized patients were offered optional VAY736 administration after week 16.
Arm/Group | VAY736 Administered at Visit 2 (Day 1) | VAY736 Administered at Visit 7 (Week 16 - Week 17) | Placebo Administered at Visit 2
Number analyzed (Participants) | 4 | 4 | 4
Participants
  On-treatment Adverse Events (AEs) | 4 | 3 | 1
  On-treatment Serious Adverse Events (SAEs) | 0 | 0 | 0
  On-treatment Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from first dosing (single administration, Day 1) up to End of Study Visit (EOS) depending on B cell recovery (ranging from week 48 to 216).
Arm/Group | VAY736 Administered at Visit 2 (Day 1) | VAY736 Administered at Visit 7 (Week 16 - Week 17) | Placebo Administered at Visit 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 Administered at Visit 2 (Day 1) (N=4) | VAY736 Administered at Visit 7 (Week 16 - Week 17) (N=4) | Placebo Administered at Visit 2 (N=4)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0
Chills (General disorders) | 2 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Glucose urine present (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 1
Hypotonia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
After enrolling 8 patients, the recruitment was terminated based on strategic considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.